CLINICAL TRIAL: NCT02377102
Title: Does Physical Therapy Prevent Total Knee Arthroplasty in Patients With End Stage Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-2152
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observational (No Intervention): Patients will be asked to continue for 12 weeks of nonoperative medical management without physical therapy. At 12 weeks they will be reevaluated regarding the need for total knee arthroplasty.
- Physical Therapy (Active Comparator): Patients will be provided a prescription for 12 weeks of physical therapy at a location of their choice. No set protocol will be issued to allow for adjustments based on patient activity level and the therapist's professional choice. The physical therapy techniques, consisting of active and passive physiological and accessory movements and soft tissue mobilization, active range of motion exercises, muscle strengthening, muscle stretching, and exercises such as riding a stationary bicycle will be applied at the discretion of the treating physical therapist primarily to the knee and surrounding structures.
  Interventions: Procedure: Physical Therapy

INTERVENTIONS:
Procedure: Physical Therapy — 12 weeks of supervised physical therapy.
  Arms: Physical Therapy

SUMMARY:
Purpose: For the target population of adult patients with end stage osteoarthritis, this randomized clinical trial will be used to evaluate the benefit of three months of physical therapy compared to no treatment in patients indicated for total knee arthroplasty.

Participants:Patients that are diagnosed with end stage osteoarthritis who are indicated for total knee arthroplasty.

Procedures: Patients will be randomized to either receive physical therapy or no treatment. They will be scheduled to return in 3 months for discussion of operative versus continued nonoperative treatment of their osteoarthritis.This will be determined by change in PROMIS (Patient Reported Outcome Measurement Information System) score and prevention of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with grade 3 and 4 (severe) osteoarthritis and indicated for primary total knee arthroplasty.

Exclusion Criteria:

* Age less than 18 y/o
* Any form of arthritis other than osteoarthritis (traumatic, rheumatic, etc)
* Previous knee surgery
* Inability to personally consent to or participate with therapy due to cognitive impairment, physical disability, intoxication or sedation
* known contraindications would include patients that will be unable to participate with therapy or who will put themselves at significant risk due to therapy (this could be either severe cardiac or respiratory impairment that prevents the patient from ambulating or mental impairment preventing the patients from following instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-02; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Prevention of surgical intervention questionnaire | 12 weeks
  Following Physical Therapy or observation, the patients (who are indicated for total knee replacement) will be asked if they desire a surgical intervention or if they would like to continue nonoperative management.

SECONDARY OUTCOMES:
PROMIS-(Patient Reported Outcomes Measurement Information System) Lower Extremity Function Score | 12 weeks
  The PROMIS score incorporates questions from multiple validated instruments of functional outcome. The system was then calibrated to the normal population distribution and has been applied previously to assess lower extremity dysfunction. This will increase our sensitivity in detecting differences between the two groups. The CAT is an adaptive test that responds to previous patient responses to decrease the amount of questions required to obtain a score. This will allow our CAT to last 1-5 minutes as opposed to a longer patient reported score or system. PROMIS has also been utilized in the setting of arthritis and should allow for a greater detection of functional improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Del Gaizo, MD, Study Director — UNC Orthopaedics
Locations (1):
- UNC Orthopaedics, Chapel Hill, North Carolina, United States